CLINICAL TRIAL: NCT04960878
Title: The Effect of Synbiotics on the Upper Respiratory Tract Infection in Healthy Subjects: A Randomized Double-Blind Trial
Brief Title: The Effect of Synbiotics on the Upper Respiratory Tract Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Liegang Liu, Professor, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2020S042
Record Dates: First submitted 2021-06-29; First posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Upper Respiratory Tract Infection; Gut Microbiota; Immune Function
MeSH Terms: conditions — Respiratory Tract Infections | interventions — Synbiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): 1.5 g maltodextrin in a sachet once daily for 8 weeks.
  Interventions: Dietary Supplement: Placebo
- Synbiotic (Experimental): 1.5 g synbiotics supplement of Lactobacillus rhamnosus HN001 (1.5×10^11 CFU) , Bifidobacterium lactis HN019 (7.5×10^10 CFU), and 500mg fructooligosaccharides in a sachet once daily for 8 weeks.
  Interventions: Dietary Supplement: Synbiotic

INTERVENTIONS:
Dietary Supplement: Synbiotic — Synbiotics sachet mainly contained Lactobacillus rhamnosus HN001, Bifidobacterium lactis HN019, and fructooligosaccharides.
  Arms: Synbiotic
Dietary Supplement: Placebo — Maltodextrin
  Arms: Placebo

SUMMARY:
Gut microbiome manipulation to alter the gut-lung axis may potentially protect humans against respiratory infections. However, clinical trials of synbiotics, one of the microbiota-targeted intervention, in this regard is few. Therefore, this study aims to examine the effect of synbiotics on the incidence and severity of upper respiratory tract infection, gut microbiota composition and function, as well as biomarkers of immune function.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-65 years；
* good general health as determined by medical questionnaires;
* BMI <35 kg/m2;

Exclusion Criteria:

* known congenital or acquired immune defects；
* allergies and other chronic or acute diseases requiring treatment；
* subjects with chronic gastrointestinal diseases;
* alcohol or drug misuse or both；
* pregnancy or lactation；
* vaccination against influenza within the last 12 months；
* use of oral antibiotics, probiotics, prebiotics, synbiotics, drugs active on gastrointestinal motility, or a laxative of any class within the last month.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2021-01-05 (Actual)

PRIMARY OUTCOMES:
The incidence of the upper respiratory tract infection | Up to 8 weeks

SECONDARY OUTCOMES:
The duration of the upper respiratory tract infection | Up to 8 weeks
The severity of the upper respiratory tract infection | Up to 8 weeks
  The severity of the upper respiratory tract infection was assessed using the 24-item Wisconsin Upper Respiratory Symptom Survey (WURSS-24). Paricipants were required to answer the question, "Did you have any symptom of upper respiratory tract infection today"? If someone answered "yes", he/she was instructed to complete WURSS-24 surveys daily.
Changes in the gut mictobiota | Baseline, 4 weeks, 8 weeks
  Changes in the composition, diversity, and function of gut mictobiota in feces will be measured by 16S rRNA gene sequencing.
Changes in the levels of sIgA in saliva and feces | Baseline, 4 weeks, 8 weeks
Changes in the levels of inflammatory cytokine | Baseline, 4 weeks, 8 weeks
  Changes in the levels of fasting plasma inflammatory cytokine, including CRP, IL-1β, IL-6, IL-8, IL-10, TNF-α, and IFN-γ.
Changes in the number of T, B, NK and monocytes populations | Baseline, 4 weeks, 8 weeks
  Changes in the number of T-lymphocytes(CD45+CD3+), B-lymphocytes(CD45+CD19+), monocytes(CD45+CD14+), and natural killer cells(CD45+CD56+) in blood samples were evaluated by flow cytometer.
Changes in the subpopulation frequencies of blood lymphocyte and dendritic cells | Baseline, 4 weeks, 8 weeks
  Changes in the subpopulation of blood lymphocytes (the levels of CD3+, CD4+, CD8+, and CD25+) and dendritic cells (the levels of CD3-CD19-CD56-HLA-DR+ CD11c+cells and CD3-CD19-CD56-HLA-DR+CD123+ cells ) in blood samples were evaluated by flow cytometer.
Change in body weight | Baseline, 4 weeks, 8 weeks
Change in BMI | Baseline, 4 weeks, 8 weeks
Change in body fat composition | Baseline, 4 weeks, 8 weeks
Change in the levels fasting plasma glucose | Baseline, 4 weeks, 8 weeks
Changes in the levels of fasting plasma TC, TG, LDL, and HDL | Baseline, 4 weeks, 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Liegang Liu, PhD, Principal Investigator — Tongji Medical College, Huazhong University of Science and Technology, Wuhan 430030, China
Locations (1):
- Huazhong University of Science and Technology, Wuhan, Hubei, China